CLINICAL TRIAL: NCT06278155
Title: Enhancing Social Relations: Training Protocol for Children With ASD
Brief Title: Social Relations Training for Children With ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2024-001
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; children; social relations; social robot; NAO
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Robotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental social relations group (Experimental): In the experimental group, a social robot is expected to mediate the relationship among peers. Its task is to prompt, reinforce and support the participants' responses. In this case, it is the therapist who mediates the relationship by prompting, reinforcing and supporting the participants' responses.
  Interventions: Other: Social relation training with social robot
- Control social relations group (Other): In the control group, the therapist is expected to act as a mediator of the relationship, prompting, reinforcing and supporting the participants' responses.
  Interventions: Other: Traditional social relations training

INTERVENTIONS:
Other: Social relation training with social robot — The protocol is divided in two sections: basic and advanced social relations.
  The "basic social relations"section consists of 4 stages:
  Stage 1 focuses on spontaneous eye contact between the child and the robot Strage 2 introduces the goal of spontaneously looking at a peer Stage 3 focuses on respecting the turn between children Stage 4 aims to encourage peer cooperation Nao social robot helps children to develop specific social skills.
  The "advanced social relation" section consists of 5 stages:
  Stage 1: The goal is to initiate physical interaction with a peer during a game Stage 2 is focused on mand (verbal requests) directed to peers Stage 3: The goal is to respond spontaneously to questions or statements from peers In the Stage 4 the child should to play with peers for at least 5 minutes Stage 5: the goal is to conduct at least 4 verbal exchanges on a given topic with peers At each stage, Nao provides verbal prompts to guide the child toward the appropriate response
  Arms: Experimental social relations group
Other: Traditional social relations training — Traditional social relations training is the same as the experimental one, however in this context the entire protocol is conducted without the aid of social robot NAO.
  Arms: Control social relations group

SUMMARY:
The following protocol was developed with the intention of significantly improving social skills by focusing on increasing relationship skills among children with ASD. Divided into two distinct parts, "Basic Social Relationships" and "Intermediate Social Relationships," the protocol has 4 stages for the former and 5 stages for the latter. Each phase is preparatory to the next, and in addition, a teaching procedure is implemented that adopts three prompt levels (partial, moderate and total), gradually aiming to reduce the assistance provided to encourage independent response. This gradual approach is designed to stimulate greater independence in social interactions.

The training lasts between 6 and 12 months, with one or two weekly group meetings lasting forty-five minutes each. Before the start and at the end of the protocol, participants are assessed using the Vineland scale to evaluate their adaptive behaviors.

The primary goal is to enable children with autism to develop meaningful social skills, providing them with concrete tools to interact more effectively and independently with their peers, thus improving their quality of life and social involvement. The protocol involves two distinct groups, experimental and control group.

The experimental group involves the use of a social robot that acts as a mediator in the interactions among participants. The role of the social robot is to facilitate, reinforce and support the participants' responses during the activities. The therapist coordinates with the social robot, helping to guide, reinforce and support participants' interactions.

In the control group, the therapist takes on the role of mediating interactions, helping and facilitating participants' responses. There is no involvement of a social robot; therefore,the therapist self acts directly to guide, reinforce and support the participants' social interactions.

ELIGIBILITY:
Inclusion Criteria:

* language in sentences
* Griffiths: QS>75

Exclusion Criteria:

* presence of other medical disorders

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
Vineland-II (Vineland Adaptive Behavior Scales-II - Survey Intervention Form) | The administration of the Vineland-II takes approximately 20-60 minutes.
  The Vineland-II, a revision of the Vineland Adaptive Behavior Scales (Vineland ABS), assess adaptive behavior (AC), i.e., the activities that the individual habitually performs to meet the expectations of personal autonomy and social responsibility characteristic of people of the same age and cultural background.
  Specifically, they aim to measure CA in the domains Communication, Skills of Daily Living, Socialization (in individuals from 0 to 90 years of age) and Motor Skills (in individuals from 0 to 7 years of age and 56 to 90 years of age). Assessment of CA is necessary for diagnosis of intellectual disability disorder and, in accordance with DSM-5, for assessment of the level of severity of the disorder.
  The Vineland-IIs consist of 4 scales divided into 11 subscales. They also provide an overall CA index.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ntaountaki, Polyxeni & Lorentzou, Georgia & Lykothanasi, Andriana & Anagnostopoulou, Panagiota & Alexandropoulou, Vasiliki & Drigas, Athanasios. (2019). Robotics in Autism Intervention. 7. 4-17. 10.3991/ijes.v7i4.11448.
- [Background] Chung, E.Yh. Robotic Intervention Program for Enhancement of Social Engagement among Children with Autism Spectrum Disorder. J Dev Phys Disabil 31, 419-434 (2019).
- [Background] Rakhymbayeva N, Amirova A, Sandygulova A. A Long-Term Engagement with a Social Robot for Autism Therapy. Front Robot AI. 2021 Jun 16;8:669972. doi: 10.3389/frobt.2021.669972. eCollection 2021. PMID 34222353